CLINICAL TRIAL: NCT00202358
Title: The Effect of Perioperative Atenolol on Post-Operative Cytokines
Brief Title: Perioperative Effect of Atenolol on Cytokine Profiles
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Saini Foundation (Other)
Collaborators: Medtronic - MITG (Industry)
Responsible Party: Vikas Saini, M.D., Cape Cod Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PEACK
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2008-06-17 (Estimated); Status verified 2008-06

CONDITIONS: Surgery
Keywords: perioperative; beta-blockers; inflammation; outcomes
MeSH Terms: conditions — Inflammation | interventions — Atenolol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- placebo (Placebo Comparator)
  Interventions: Drug: placebo
- atenolol (Experimental)
  Interventions: Drug: atenolol

INTERVENTIONS:
Drug: atenolol
  Arms: atenolol
Drug: placebo
  Arms: placebo

SUMMARY:
Studies have shown that beta-blockers such as atenolol when given in the perioperative period reduce morbidity and mortality. One study showed that atenolol given just during the surgery period, seemed to improve outcomes up to 2 years later. This is hard to explain since beta-blockers act on the body by blocking the effects of adrenalin and thereby lowering heart rate and blood pressure.

This study is designed to find out if perioperative atenolol might exert its long term effects through an anti-inflammatory mechanism rather than by lowering heart rate and blood pressure. It is known that inflammation increases after surgery as part of the healing process. However, it is also becoming clear that low-grade chronic inflammation can also lead to long term adverse effects.

ELIGIBILITY:
Inclusion Criteria:

* elective abdominal, orthopedic, or gynecologic surgery
* ability to give informed consent
* ability to tolerate beta-blocker therapy
* ability to comply with follow-up requirements

Exclusion Criteria:

* currently receiving beta-blocker therapy
* EKG documented 2nd or 3rd degree heart block
* EKG documented sinus bradycardia
* Serum creatinine > 2.0
* current treatment asthma
* history of rheumatoid arthritis
* history of Crohn's disease
* history of lupus
* history of inflammatory cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2002-11; Primary Completion 2007-11 (Actual); Study Completion 2008-09 (Estimated)

PRIMARY OUTCOMES:
Postoperative levels of IL-6 and C-Reactive protein | 6 hrs, 48 hrs, 6 weeks

SECONDARY OUTCOMES:
IL-10, TNF-α | 6 hrs, 48 hrs, 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Vikas Saini, M.D., Principal Investigator — Dept Medicine, Cape Cod Hospital
Locations (1):
- Cape Cod Hospital, Hyannis, Massachusetts, United States